CLINICAL TRIAL: NCT00472381
Title: Assessment of Continuous Intravenous Insulin Protocol Versus Subcutaneous Insulin in Acute Ischemic Stroke
Brief Title: Efficacy and Safety of Continuous Intravenous Versus Usual Subcutaneous Insulin in Acute Ischemic Stroke
Acronym: INSULINFARCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060202
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2012-09

CONDITIONS: Acute Stroke; Acute Cerebral Ischemia
Keywords: Acute Ischemic Stroke; Post-Stroke Hyperglycaemia; Insulin treatment; Insulin; DWI; MRI
MeSH Terms: conditions — Stroke; Ischemic Stroke; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Experimental): Insulin
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin

SUMMARY:
Hyperglycaemia is a frequent finding in acute ischemic stroke and associated with poor outcome. But the modalities of glucose lowering are still debated. This study will test the efficacy and safety of continuous intravenous insulin protocol versus usual subcutaneous insulin in acute ischemic stroke.

DETAILED DESCRIPTION:
It is demonstrated that post-stroke hyperglycaemia is associated with poor outcome. Yet, the efficiency of aggressive insulin serum glucose control is not established. Furthermore the modalities of insulin administration are discussed since US and European guidelines recommend subcutaneous administration, whereas some groups use intravenous administration of insulin. The purpose of this study is to compare the efficacy and the safety of a continuous intravenous insulin protocol versus classical subcutaneous administration of insulin. The study will include carotid territory stroke at the acute stage (< 6 hours of onset) confirmed by MRI, and randomized in intravenous versus subcutaneous insulin. The percentage of patients in the target range (mean capillary glycaemia within 24 hours < 7 mmol/l) is the primary outcome. The secondary outcomes include comparison of Modified Rankin Scale at 3 months, rate of hypoglycaemic events and comparison of Infarct Growth as measured on MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Carotid territory stroke
* MRI performed in the first five hours of stroke onset
* Baseline National Institutes of Health Stroke Scale (NIHSS) > 4 or < 26
* Time between MRI and treatment under one hour

Exclusion Criteria:

* Pre-existing Modified Rankin Scale of three or higher
* Advanced or terminal illness with risk of death in the next 6 months, addiction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in the glucose target range within 24 hours of the initiation of treatment. | 24 hours

SECONDARY OUTCOMES:
Modified Rankin Scale at three months | three months
Magnetic resonance imaging (MRI) infarct growth at one day | one day
Percentage of patients with hypoglycaemic event (< 3 mmol/l) | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Yves Samson, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- AP-HP Urgences cerebro vasculaires La Pitié Salpétrière, Poissy, France

REFERENCES:
- [Result] Samson Y, Bruandet M, Lejeune M, Deltour S, Grimaldi A. [Insulin in the treatment of ischemic stroke]. Presse Med. 2006 Apr;35(4 Pt 2):696-8. doi: 10.1016/s0755-4982(06)74664-4. French. PMID 16614616
- [Derived] Rosso C, Pires C, Corvol JC, Baronnet F, Crozier S, Leger A, Deltour S, Valabregue R, Amor-Sahli M, Lehericy S, Dormont D, Samson Y. Hyperglycaemia, insulin therapy and critical penumbral regions for prognosis in acute stroke: further insights from the INSULINFARCT trial. PLoS One. 2015 Mar 20;10(3):e0120230. doi: 10.1371/journal.pone.0120230. eCollection 2015. PMID 25793765
- [Derived] Rosso C, Corvol JC, Pires C, Crozier S, Attal Y, Jacqueminet S, Deltour S, Multlu G, Leger A, Meresse I, Payan C, Dormont D, Samson Y. Intensive versus subcutaneous insulin in patients with hyperacute stroke: results from the randomized INSULINFARCT trial. Stroke. 2012 Sep;43(9):2343-9. doi: 10.1161/STROKEAHA.112.657122. Epub 2012 Jun 14. PMID 22700528
- See also: DOI:10.1161/STROKEAHA.112.657122 — http://stroke.ahajournals.org